CLINICAL TRIAL: NCT03047395
Title: A Multicenter, Open Label Study to Assess the Safety and Efficacy of Risankizumab for Maintenance in Moderate to Severe Plaque Type Psoriasis (LIMMITLESS)
Brief Title: A Study to Assess the Safety and Efficacy of Risankizumab for Maintenance in Moderate to Severe Plaque Type Psoriasis ( LIMMITLESS )
Acronym: LIMMITLESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-997; 2016-003046-87 (EudraCT Number); 1311.31 (Other: AbbVie)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Risankizumab (Experimental): Participants will receive risankizumab administered by subcutaneous injection.
  Interventions: Biological: risankizumab

INTERVENTIONS:
Biological: risankizumab — Risankizumab 150 mg administered by subcutaneous injection every 12 weeks.
  Other Names: ABBV-066; Skyrizi; BI 655066

SUMMARY:
The purpose of this study is to investigate the long-term safety and efficacy of risankizumab in the treatment of moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
This is a Phase 3, single-arm, multicenter open label extension (OLE) study designed to investigate the long-term safety and efficacy of 150 mg risankizumab in the treatment of moderate to severe chronic plaque psoriasis. Approximately 2200 participants who meet the entry criteria are planned to be enrolled in this study, rolling over from the preceding Phase 2/3 studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of moderate to severe chronic plaque psoriasis, who have completed one of the preceding studies.
* Participants must be candidates for prolonged open label risankizumab treatment according to investigator judgment.
* Females of childbearing potential must have a negative urine pregnancy test result at Baseline.

If female, participant must be either postmenopausal, OR permanently surgically sterile OR for women of childbearing potential practicing at least one protocol specified method of birth control, starting at Baseline through at least 20 weeks after the last dose of study drug.

- Participants must have signed and dated a written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission into the study.

Exclusion Criteria:

* Premature discontinuation for any reason in the preceding study.
* Participants who have developed guttate, erythrodermic, pustular or drug-induced psoriasis as diagnosed by the investigator during the preceding study.
* Use of any prohibited medication or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator.
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and ECG), or laboratory value outside the reference range that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the study, compromise the safety of the subject, or compromise the quality of the data.
* Previous enrollment in this study.
* Female subject who is pregnant, breastfeeding or is considering becoming pregnant during the study or within 20 weeks after the last dose of study drug.
* Time elapsed is > 8 weeks since the completion visit in the preceding study.
* Participant is considered by the investigator for any reason, to be an unsuitable candidate for the study and not able to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2170 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (233):
- United States (79):
  - Total Skin and Beauty Dermatology Center /ID# 154000, Birmingham, Alabama
  - University of Alabama at Birmingham - Main /ID# 153983, Birmingham, Alabama
  - NW Arkansas Clinical Trials Center /ID# 154014, Rogers, Arkansas
  - Bakersfield Derma & Skin Cance /ID# 154008, Bakersfield, California
  - California Dermatology and Research Institute /ID# 154007, Encinitas, California
  - T. Joseph Raoof, MD, Inc. /ID# 154078, Encino, California
  - Center for Dermatology Clinical Research /ID# 154009, Fremont, California
  - Kaiser Permanente Los Angeles /ID# 154079, Los Angeles, California
  - Dermatology Research Associates /ID# 153977, Los Angeles, California
  - Wallace Medical Group /ID# 154025, Los Angeles, California
  - Dermatology Specialists, Inc /ID# 153984, Oceanside, California
  - Huntington Medical Foundation /ID# 154002, Pasadena, California
  - Medderm Associates /ID# 154098, San Diego, California
  - Southern California Dermatology /ID# 154006, Santa Ana, California
  - UNISON Center for Clinical Tri /ID# 153979, Sherman Oaks, California
  - New England Research Associates, LLC /ID# 154004, Bridgeport, Connecticut
  - UConn Health /ID# 154128, Farmington, Connecticut
  - Florida Academic Centers Research /ID# 154045, Coral Gables, Florida
  - Leavitt Medical Associates of Florida /ID# 154046, Ormond Beach, Florida
  - Progressive Medical Research /ID# 154027, Port Orange, Florida
  - Hamilton Research, LLC /ID# 153980, Alpharetta, Georgia
  - Advanced Medical Research, PC /ID# 153999, Sandy Springs, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 153974, Chicago, Illinois
  - Rush University Medical Center /ID# 154099, Chicago, Illinois
  - Arlington Dermatology /ID# 153975, Rolling Meadows, Illinois
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 154011, Skokie, Illinois
  - Dundee Dermatology /ID# 154110, West Dundee, Illinois
  - Dawes Fretzin, LLC /ID# 154146, Indianapolis, Indiana
  - The Dermatology Center PSC - New Albany /ID# 154075, New Albany, Indiana
  - The Indiana Clinical Trials Center /ID# 153976, Plainfield, Indiana
  - The South Bend Clinic Center /ID# 154147, South Bend, Indiana
  - Epiphany Dermatology of Kansas LLC /ID# 153993, Overland Park, Kansas
  - Skin Sciences, PLLC /ID# 153991, Louisville, Kentucky
  - DS Research /ID# 154028, Louisville, Kentucky
  - Massachusetts General Hospital /ID# 153990, Boston, Massachusetts
  - ActivMed Practices and Research, LLC. /ID# 154044, Methuen, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 154111, Ann Arbor, Michigan
  - Great Lakes Research Group - Bay City /ID# 153998, Bay City, Michigan
  - Michigan Center for Skin Care Research /ID# 153986, Clinton Township, Michigan
  - Somerset Skin Centre /ID# 154097, Troy, Michigan
  - Minnesota Clinical Study Center /ID# 154015, New Brighton, Minnesota
  - Central Dermatology, PC /ID# 154013, St Louis, Missouri
  - Skin Specialists, PC /ID# 154024, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 154095, Lebanon, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey /ID# 154001, East Windsor, New Jersey
  - Schweiger Dermatology Group /ID# 202489, Verona, New Jersey
  - Forest Hills Dermatology Group /ID# 154113, Kew Gardens, New York
  - Icahn School of Medicine at Mount Sinai /ID# 154129, New York, New York
  - The Rockefeller University /ID# 153994, New York, New York
  - DermResearchCenter of New York, Inc. /ID# 154012, Stony Brook, New York
  - Buffalo Medical Group /ID# 154148, Williamsville, New York
  - Darst Dermatology /ID# 154076, Charlotte, North Carolina
  - Dermatology Consulting Service /ID# 154010, High Point, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 202490, Raleigh, North Carolina
  - Wilmington Dermatology Center /ID# 154109, Wilmington, North Carolina
  - Synexus Research Cincinnati /ID# 153997, Cincinnati, Ohio
  - Oregon Dermatology and Research Center /ID# 153982, Portland, Oregon
  - Oregon Medical Research Center /ID# 154003, Portland, Oregon
  - Altoona Ctr Clinical Res /ID# 153981, Duncansville, Pennsylvania
  - Paddington Testing Co., Inc. /ID# 154022, Philadelphia, Pennsylvania
  - University of Pittsburgh MC /ID# 153995, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC /ID# 154096, Johnston, Rhode Island
  - Coastal Clinical Research Center of the Carolinas /ID# 154112, Charleston, South Carolina
  - Synexus Clinical Research US, Inc. /ID# 154127, Greer, South Carolina
  - Coastal Carolina Research Center /ID# 153992, North Charleston, South Carolina
  - Health Concepts /ID# 153996, Rapid City, South Dakota
  - Austin Dermatology Associates /ID# 154042, Austin, Texas
  - Bellaire Dermatology Associates /ID# 153987, Bellaire, Texas
  - Modern Research Associates, PLLC /ID# 154043, Dallas, Texas
  - Menter Dermatology Res Inst /ID# 153985, Dallas, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 154005, Houston, Texas
  - Suzanne Bruce and Associates-Houston /ID# 154026, Houston, Texas
  - Derm Clin Res Ctr San Antonio /ID# 153978, San Antonio, Texas
  - Progressive Clinical Research /ID# 154149, San Antonio, Texas
  - Dermatology San Antonio /ID# 154077, San Antonio, Texas
  - Center for Clinical Studies Webster TX /ID# 154150, Webster, Texas
  - Virginia Clinical Research, Inc. /ID# 154016, Norfolk, Virginia
  - Dermatology Associates of Seattle /ID# 153988, Seattle, Washington
  - Premier Clinical Research /ID# 154284, Spokane, Washington
- Australia (7):
  - Paratus Clinical Research Woden /ID# 154307, Phillip, Australian Capital Territory
  - St George Dermatology & Skin Cancer Centre /ID# 154308, Kogarah, New South Wales
  - Specialist Connect Pty Ltd /ID# 154311, Woolloongabba, Queensland
  - North Eastern Health Specialists /ID# 154309, Campbelltown, South Australia
  - Skin Health Institute Inc /ID# 154305, Carlton, Victoria
  - Sinclair Dermatology - Melbourne /ID# 154310, Melbourne, Victoria
  - Fremantle Dermatology /ID# 154306, Fremantle, Western Australia
- Austria (3):
  - Klinik Landstrasse /ID# 154300, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 154302, Vienna, Vienna
  - Landeskrankenhaus Feldkirch /ID# 154303, Feldkirch, Vorarlberg
- Belgium (6):
  - Cliniques Universitaires de Bruxelles Hopital Erasme /ID# 154293, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 154295, Jette, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 154294, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege Sart Tilman /ID# 154297, Liège, Liege
  - UZ Gent /ID# 154296, Ghent, Oost-Vlaanderen
  - IMTR - Grand Hopital de Charleroi /ID# 154298, Loverval
- Canada (26):
  - Kirk Barber Research, CA /ID# 153840, Calgary, Alberta
  - Dermatology Research Institute Inc. /ID# 153850, Calgary, Alberta
  - Stratica Medical /ID# 153848, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 153842, Surrey, British Columbia
  - Enverus Medical Research /ID# 153851, Surrey, British Columbia
  - Karma Clinical Trials /ID# 153876, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Resea /ID# 153870, Halifax, Nova Scotia
  - CCA Medical Research /ID# 153859, Ajax, Ontario
  - Kingsway Clinical Research /ID# 154292, Etobicoke, Ontario
  - Dermatrials Research /ID# 153847, Hamilton, Ontario
  - The Guenther Dermatology Research Centre /ID# 153841, London, Ontario
  - Lynderm Research Inc. /ID# 153861, Markham, Ontario
  - DermEdge Research Inc. /ID# 153843, Mississauga, Ontario
  - North Bay Dermatology Centre /ID# 153845, North Bay, Ontario
  - The Centre for Clinical Trials /ID# 153871, Oakville, Ontario
  - Dermatology Ottawa Research Centre /ID# 153862, Ottawa, Ontario
  - SKiN Centre for Dermatology /ID# 153853, Peterborough, Ontario
  - The Center For Dermatology /ID# 153844, Richmond Hill, Ontario
  - York Dermatology Clinic and Research Centre /ID# 153860, Richmond Hill, Ontario
  - Toronto Research Centre /ID# 153852, Toronto, Ontario
  - Research Toronto /ID# 153854, Toronto, Ontario
  - K. Papp Clinical Research /ID# 153855, Waterloo, Ontario
  - XLR8 Medical Research /ID# 153858, Windsor, Ontario
  - Windsor Clinical Research, Inc /ID# 153877, Windsor, Ontario
  - Innovaderm Research Inc. /ID# 153846, Montreal, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 153856, Québec, Quebec
- Czechia (6):
  - DERMAMEDICA, s.r.o. /ID# 153890, Červený Kostelec
  - Medical research s.r.o. /ID# 153898, Ostrava
  - Clintrial s.r.o. /ID# 153889, Prague
  - MUDr. Blanka Havlickova - dermatovenerologie /ID# 153888, Prague
  - Pratia Prague s.r.o. /ID# 153897, Prague
  - CCR Czech a.s /ID# 153887, Prague
- Finland (2):
  - Terveystalo Tampere /ID# 154118, Tampere
  - Mehilainen Turku /ID# 154120, Turku
- France (3):
  - Chu de Nice-Hopital Larchet Ii /Id# 153948, Nice, Alpes-Maritimes
  - Hôpital Charles-Nicolle /ID# 205842, Rouen
  - CHU Toulouse - Hopital Larrey /ID# 153951, Toulouse
- Germany (25):
  - Universitaetsklinik Heidelberg /ID# 153910, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 153912, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 154093, Erlangen, Bavaria
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 153892, Blankenfelde-Mahlow, Brandenburg
  - Klinikum Darmstadt GmbH /ID# 153893, Darmstadt, Hesse
  - Universitaetsklinikum Frankfurt /ID# 153891, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 153895, Munster, Lower Saxony
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 154092, Mainz, Rhineland-Palatinate
  - CMS3 Company for Medical Study /ID# 201318, Selters, Rhineland-Palatinate
  - Universitaetsklinikum Leipzig /ID# 153909, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 153916, Kiel, Schleswig-Holstein
  - DermaKiel Allergie und Haut Centrum /ID# 201316, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 153896, Berlin
  - ISA Interdisciplinary Study Association GmbH /ID# 153907, Berlin
  - Hautarztpraxis Dr. Niesmann und Dr. Othlinghaus /ID# 154289, Bochum
  - Universitaetsklinikum Bonn /ID# 154094, Bonn
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 153906, Dresden
  - Universitaetsmedizin Goettingen /ID# 154091, Göttingen
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 154089, Hamburg
  - Klinische Forschung Hamburg GmbH /ID# 154290, Hamburg
  - TFS Trial Form Support GmbH /ID# 153894, Hamburg
  - Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 153915, Munich
  - Klinische Forschung Schwerin GmbH /ID# 154291, Schwerin
  - Hautarztpraxis Dr. med. Matthias Hoffmann /ID# 153917, Witten
  - CentroDerm GmbH /ID# 153914, Wuppertal
- Japan (39):
  - Nagoya City University Hospital /ID# 153866, Nagoya, Aichi-ken
  - Fukuoka University Hospital /ID# 153864, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 156320, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 153873, Fukushima, Fukushima
  - Gifu University Hospital /ID# 169410, Gifu, Gifu
  - JR Sapporo Hospital /ID# 201963, Sapporo, Hokkaido
  - Medical Corporation Kojinkai Sapporo Skin Clinic /ID# 154083, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 154285, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 170706, Kobe, Hyōgo
  - Iwate Medical University Hospital /ID# 170843, Shiwa-gun, Iwate
  - Kagawa University Hospital /ID# 168656, Kita-gun, Kagawa-ken
  - Japan Organization of Occupational Health and Society Kanto Rosai Hospital /ID# 169172, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 153867, Sagamihara-shi, Kanagawa
  - Yokohama City University Hospital /ID# 168831, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 169415, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 156318, Kyoto, Kyoto
  - Mie University Hospital /ID# 156317, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 169006, Sendai, Miyagi
  - Shinshu University Hospital /ID# 170937, Matsumoto-shi, Nagano
  - Nagasaki University Hospital /ID# 170219, Nagasaki, Nagasaki
  - Okayama University Hospital /ID# 200631, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 170884, Hirakata-shi, Osaka
  - Osaka Metropolitan University Hospital /ID# 153869, Osaka, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 156319, Osaka, Osaka
  - Kindai University Hospital /ID# 153865, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 156321, Suita-shi, Osaka
  - Hamamatsu University Hospital /ID# 170132, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital /ID# 154286, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital /ID# 200292, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 154084, Bunkyo-ku, Tokyo
  - Tokyo Teishin Hospital /ID# 165912, Chiyoda-ku, Tokyo
  - St.Luke's International Hospital /ID# 153863, Chuo-ku, Tokyo
  - Teikyo University Hospital /ID# 154287, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital /ID# 154081, Itabashi-ku, Tokyo
  - The Jikei University Hospital /ID# 154080, Minato-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 154082, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 153874, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 153868, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital /ID# 156322, Ube-shi, Yamaguchi
- Mexico (3):
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 153882, Monterrey, Nuevo León
  - Derma Norte del Bajio S.C. /ID# 153880, Aguascalientes
  - Centro de Dermatologia de Monterrey /ID# 153881, Monterrey
- Poland (10):
  - Solumed Centrum Medyczne /ID# 153466, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow /ID# 153472, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocawiu /ID# 153473, Wroclaw, Lower Silesian Voivodeship
  - KO-MED Centra Kliniczne Lublin /ID# 153469, Lublin, Lublin Voivodeship
  - High-Med Przychodnia Specjalistyczna /ID# 153468, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 153467, Warsaw, Masovian Voivodeship
  - Osteo-Medic S.C. /ID# 156535, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne /ID# 153471, Gdansk, Pomeranian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 153884, Gdansk, Pomeranian Voivodeship
  - Dermoklinika Medical Center /ID# 153470, Lodz, Łódź Voivodeship
- Portugal (4):
  - 2CA-Braga, Hospital de Braga /ID# 156323, Braga
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 153462, Lisbon
  - CHP, EPE- Hospital Geral de Sa /ID# 153464, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 153463, Porto
- South Korea (9):
  - Gachon University Gil Medical Center /ID# 153489, Incheon, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 153491, Seongnam, Gyeonggido
  - Chonnam National University Hospital /ID# 153488, Gwangju, Jeonranamdo
  - KonKuk University Medical Center /ID# 153483, Seoul, Seoul Teugbyeolsi
  - Korea Universtiy Guro Hospital /ID# 153490, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital /ID# 153486, 서초구, Seoul Teugbyeolsi
  - Pusan National University Hospital /ID# 153485, Busan
  - Seoul National University Hospital /ID# 153484, Seoul
  - Samsung Medical Center /ID# 153487, Seoul
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol /ID# 153465, Badalona, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 154125, Barcelona
  - Hospital Universitario Infanta Leonor /ID# 154121, Madrid
  - Hospital General Universitario de Valencia /ID# 154126, Valencia
- Sweden (3):
  - Karolinska University Hospital Solna /ID# 154131, Solna, Stockholm County
  - Sahlgrenska University Hospital /ID# 154132, Gothenburg, Västra Götaland County
  - Sodersjukhuset /ID# 154130, Stockholm
- Taiwan (4):
  - National Taiwan University Hospital /ID# 154136, Taipei City, Taipei
  - Taipei Medical University Shuang Ho Hospital /ID# 154134, New Taipei City
  - National Cheng Kung University Hospital /ID# 154135, Tainan
  - Taiwan Adventist Hospital /ID# 154137, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Papp KA, Lebwohl MG, Puig L, Ohtsuki M, Beissert S, Gooderham M, Amin AZ, Wu T, Rubant S, Bialik B, Ashley D, Soliman AM, Chen MM, Blauvelt A. Long-Term Safety and Efficacy of Risankizumab to Treat Moderate-to-Severe Plaque Psoriasis: Final LIMMitless Phase 3, Open-Label Extension Trial Results. Am J Clin Dermatol. 2025 Sep;26(5):829-841. doi: 10.1007/s40257-025-00964-6. Epub 2025 Jul 29. PMID 40728772
- [Derived] Alexis AF, Gooderham M, Kwatra SG, Amin A, Taylor S, Espaillat R, Rettig T, Wu T, Shi L, Kaldas MI, Dilley DM, Sinvhal R, Nduaka C, Lockshin B. A Descriptive, Post Hoc Analysis of Efficacy and Safety of Risankizumab in Diverse Racial and Ethnic Patient Populations With Moderate-to-Severe Psoriasis. Dermatol Ther (Heidelb). 2024 Oct;14(10):2877-2887. doi: 10.1007/s13555-024-01268-z. Epub 2024 Oct 2. PMID 39358667
- [Derived] Hsieh CY, Hsu FL, Tsai TF. Comparison of Drug-Free Remission after the End of Phase III Trials of Three Different Anti-IL-23 Inhibitors in Psoriasis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2607-2620. doi: 10.1007/s13555-024-01229-6. Epub 2024 Jul 29. PMID 39073712
- [Derived] Papp KA, Lebwohl MG, Puig L, Ohtsuki M, Beissert S, Zeng J, Rubant S, Sinvhal R, Zhao Y, Soliman AM, Alperovich G, Leonardi C. Long-term efficacy and safety of risankizumab for the treatment of moderate-to-severe plaque psoriasis: interim analysis of the LIMMitless open-label extension trial beyond 3 years of follow-up. Br J Dermatol. 2021 Dec;185(6):1135-1145. doi: 10.1111/bjd.20595. Epub 2021 Sep 21. PMID 34157132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from Studies M16-008 (NCT02684370), M16-010 (NCT02694523), M15-995 (NCT02684357), M16-178 (NCT03255382), M16-009 (NCT02203851), M15-992 (NCT02672852), and M16-004 (NCT03000075) entered this open-label extension (OLE) study from 232 sites across 17 countries (Australia, Austria, Belgium, Canada, Czech Republic, Finland, France, Germany, Japan, Mexico, Poland, Portugal, Republic of Korea, Spain, Sweden, Taiwan, and US).
Groups:
- Risankizumab 150 mg: Risankizumab 150 mg administered by subcutaneous injection every 12 weeks.
Period: Overall Study
Arm/Group | Risankizumab 150 mg
Started | 2170
Completed | 1601 (Two of these participants completed the study but did not fill out the study completion forms.)
Not Completed | 569
Not completed — Adverse Event | 142
Not completed — Withdrawal by Subject | 155
Not completed — Lost to Follow-up | 144
Not completed — COVID-19 Infection | 2
Not completed — COVID-19 Logistical Restrictions | 9
Not completed — Other, Not Specified | 117

BASELINE CHARACTERISTICS:
Arm/Group | Risankizumab 150 mg
Number analyzed (Participants) | 2170
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 658
  40 - < 65 years | 1264
  >= 65 years | 248
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 634
  Male | 1536
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 257
  Not Hispanic or Latino | 1913
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15
  Asian | 466
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 50
  White | 1622
  More than one race | 8
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events and Non-Serious Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Median follow-up time of 1905 days
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab 150 mg
Number analyzed (Participants) | 2170
Participants
  Serious Adverse Events | 435
  Non-serious Adverse Events | 1215

ADVERSE EVENTS:
Time Frame: Median follow-up time of 1905 days
Arm/Group | Risankizumab 150 mg
All-Cause Mortality (participants affected / at risk) | 28/2170
Serious Adverse Events (participants affected / at risk) | 435/2170
Other Adverse Events (participants affected / at risk) | 1215/2170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 150 mg (N=2170)
ANAEMIA (Blood and lymphatic system disorders) | 3 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 13 (13)
ANGINA PECTORIS (Cardiac disorders) | 2 (2)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 9 (9)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 2 (2)
BIFASCICULAR BLOCK (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 (6)
CARDIAC VENTRICULAR THROMBOSIS (Cardiac disorders) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 9 (9)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 (1)
DRESSLER'S SYNDROME (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 9 (9)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1)
CONGENITAL CYSTIC KIDNEY DISEASE (Congenital, familial and genetic disorders) | 1 (1)
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1 (1)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 2 (2)
GOITRE (Endocrine disorders) | 1 (1)
GRAVES' DISEASE (Endocrine disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 (1)
THYROTOXIC CRISIS (Endocrine disorders) | 1 (1)
BLINDNESS UNILATERAL (Eye disorders) | 1 (1)
CATARACT (Eye disorders) | 3 (4)
EPIRETINAL MEMBRANE (Eye disorders) | 2 (2)
MACULAR HOLE (Eye disorders) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1)
ABDOMINAL INCARCERATED HERNIA (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 3 (3)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (2)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (2)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (2)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
RECTAL STENOSIS (Gastrointestinal disorders) | 1 (1)
RETROPERITONEAL MASS (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2)
TOOTH DISORDER (Gastrointestinal disorders) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 6 (6)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1)
SUDDEN DEATH (General disorders) | 1 (1)
SURGICAL FAILURE (General disorders) | 1 (1)
VASCULAR STENT STENOSIS (General disorders) | 1 (1)
ALCOHOLIC LIVER DISEASE (Hepatobiliary disorders) | 1 (1)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4 (5)
CHOLELITHIASIS (Hepatobiliary disorders) | 6 (6)
CIRRHOSIS ALCOHOLIC (Hepatobiliary disorders) | 1 (1)
GALLBLADDER POLYP (Hepatobiliary disorders) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 4 (4)
HEPATITIS ALCOHOLIC (Hepatobiliary disorders) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
ABSCESS JAW (Infections and infestations) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 2 (3)
APPENDICITIS (Infections and infestations) | 6 (6)
ARTHRITIS BACTERIAL (Infections and infestations) | 3 (3)
BRONCHIOLITIS (Infections and infestations) | 1 (1)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 13 (14)
COVID-19 PNEUMONIA (Infections and infestations) | 7 (7)
CELLULITIS (Infections and infestations) | 5 (6)
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 1 (1)
CHRONIC TONSILLITIS (Infections and infestations) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 6 (6)
EPIDIDYMITIS (Infections and infestations) | 1 (2)
ERYSIPELAS (Infections and infestations) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FALLOPIAN TUBE ABSCESS (Infections and infestations) | 1 (1)
FOURNIER'S GANGRENE (Infections and infestations) | 1 (1)
GAS GANGRENE (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 2 (2)
INFECTIVE GLOSSITIS (Infections and infestations) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1)
LARGE INTESTINE INFECTION (Infections and infestations) | 1 (1)
MEDIASTINAL ABSCESS (Infections and infestations) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
NEUROSYPHILIS (Infections and infestations) | 1 (1)
ORCHITIS (Infections and infestations) | 2 (3)
OSTEOMYELITIS (Infections and infestations) | 4 (4)
PERICORONITIS (Infections and infestations) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1)
PERITONITIS (Infections and infestations) | 2 (2)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 7 (7)
PNEUMONIA ASPIRATION (Infections and infestations) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1)
PSOAS ABSCESS (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 3 (3)
PYELONEPHRITIS ACUTE (Infections and infestations) | 2 (3)
RENAL ABSCESS (Infections and infestations) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 6 (6)
SEPTIC SHOCK (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 2 (2)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 (1)
COLON INJURY (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1)
CRANIOFACIAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 (2)
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 2 (2)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 2 (2)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 2 (2)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1)
NAIL INJURY (Injury, poisoning and procedural complications) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 (2)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
TENDON DISLOCATION (Injury, poisoning and procedural complications) | 2 (2)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 2 (2)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 (3)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 (2)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 6 (6)
LOOSE BODY IN JOINT (Musculoskeletal and connective tissue disorders) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 17 (20)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 3 (3)
SPINAL LIGAMENT OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 4 (4)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1)
TENDINOUS CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BORDERLINE MUCINOUS TUMOUR OF OVARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CHROMOPHOBE RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ENDOMETRIAL CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GERM CELL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
INVASIVE LOBULAR BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LARYNGEAL CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LIPOSARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
PANCREATIC CARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PENILE SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SARCOMA UTERUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SCHWANNOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SUPERFICIAL SPREADING MELANOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TRIPLE NEGATIVE BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE MYOMA EXPULSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BELL'S PALSY (Nervous system disorders) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 4 (4)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 5 (5)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 (3)
DEMENTIA (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 5 (5)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 2 (2)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PROGRESSIVE SUPRANUCLEAR PALSY (Nervous system disorders) | 1 (1)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SENSORY DISTURBANCE (Nervous system disorders) | 1 (1)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 7 (7)
THALAMIC INFARCTION (Nervous system disorders) | 2 (2)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 5 (5)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 3 (3)
ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 2 (2)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 2 (2)
ANOREXIA NERVOSA (Psychiatric disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 2 (2)
CATATONIA (Psychiatric disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 3 (4)
POST-TRAUMATIC AMNESTIC DISORDER (Psychiatric disorders) | 1 (1)
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1)
SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
CALCULUS URINARY (Renal and urinary disorders) | 2 (2)
CYSTITIS INTERSTITIAL (Renal and urinary disorders) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 8 (9)
PELVI-URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 (1)
PYELOCALIECTASIS (Renal and urinary disorders) | 1 (1)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
RENAL CYST (Renal and urinary disorders) | 1 (1)
BALANOPOSTHITIS (Reproductive system and breast disorders) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
BREAST ENLARGEMENT (Reproductive system and breast disorders) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1)
ENDOMETRIAL DISORDER (Reproductive system and breast disorders) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 1 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 (7)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 2 (2)
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 1 (1)
PRECANCEROUS SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2)
LOSS OF PERSONAL INDEPENDENCE IN DAILY ACTIVITIES (Social circumstances) | 1 (1)
ABDOMINOPLASTY (Surgical and medical procedures) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 4 (4)
AORTIC ANEURYSM (Vascular disorders) | 3 (3)
AORTIC STENOSIS (Vascular disorders) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
EMBOLISM ARTERIAL (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2)
HYPERTENSIVE URGENCY (Vascular disorders) | 1 (1)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 1 (1)
VASCULAR STENOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 150 mg (N=2170)
COVID-19 (Infections and infestations) | 360 (384)
NASOPHARYNGITIS (Infections and infestations) | 480 (833)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 312 (467)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 217 (267)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 124 (142)
HEADACHE (Nervous system disorders) | 134 (211)
HYPERTENSION (Vascular disorders) | 227 (245)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03047395/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03047395/SAP_001.pdf